CLINICAL TRIAL: NCT01828788
Title: Postoperative Rehabilitation After Cardiac Surgery in Patients at Risk of Respiratory Complications. Effects of a Continuous Bi-laterosternal Infusion of Ropivacaine Through Multihole Catheters.
Acronym: BLS-Sterno
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHU-0151
Record Dates: First submitted 2013-04-02; First posted 2013-04-11 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Scheduled Cardiac Surgery; Sternotomy; Elderly Patients; Obesity; Chronic Bronchitis
Keywords: Sternotomy; Anesthesia; Post-operative pain
MeSH Terms: conditions — Obesity; Bronchitis, Chronic; Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Ropivacaïne (Experimental): Prospective, controlled, randomised, parallel, single-centre, single-blinded trial, comparing to a control (conventional care with no locoregional anaesthesia) an infusion of ropivacaine through two multihole catheters placed lateral to the sternum. In both groups, postoperative analgesia will be achieved by paracetamol plus titrated then self-administered intravenous morphine.
  Interventions: Drug: Ropivacaine
- Placebo (Placebo Comparator): Prospective, controlled, randomised, parallel, single-centre, single-blinded trial, comparing to a control (conventional care with no locoregional anaesthesia) an infusion of ropivacaine through two multihole catheters placed lateral to the sternum. In both groups, postoperative analgesia will be achieved by paracetamol plus titrated then self-administered intravenous morphine.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Ropivacaine
  Arms: Ropivacaïne
Drug: placebo
  Arms: Placebo

SUMMARY:
Postoperative pain after cardiac surgery is a risk factor for postoperative complications. In cardiac surgery, pain is more intense during the first 48 hours and disturbs the patient's capacity of coughing, deep breathing, and early mobilisation. It may be responsible for respiratory complications such as bronchial or pulmonary infection, and may also delay the patient's rehabilitation and therefore prolong the duration of in-hospital stay. A previous pilot study performed in our department showed a sensible improvement of analgesia at movement and of rehabilitation with a continuous bilaterosternal infusion of local anaesthesia [Eljezi et al.. Reg Anesth Pain Med 2012; 37:166]. Such strategy shall be tested in a subpopulation of patients at risk for respiratory complication.

DETAILED DESCRIPTION:
Prospective, controlled, randomised, parallel, single-centre, single-blinded trial, comparing to a control (conventional care with no locoregional anaesthesia) an infusion of ropivacaine through two multihole catheters placed lateral to the sternum. In both groups, postoperative analgesia will be achieved by paracetamol plus titrated then self-administered intravenous morphine.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled cardiac surgery (aortic or mitral valve replacement, or coronary bypass surgery) with sternotomy.
* Patients will be at risk of noncardiac postoperative complications, i.e. age over 75, BMI over 30, pulmonary disease, or active smoking habit

Exclusion Criteria:

* surgery in emergency
* thoracotomy
* cardiac graft
* redo
* aortic dissection
* age over 85
* pregnancy
* patient's refusal
* minor or adult under legal protection
* psychiatric ongoing disease
* addiction to opiates
* ongoing opiate treatment
* inability to use a PCA device
* respiratory insufficiency (Vital capacity or maximal expired volume per sec. < 50% of the expected value, or mean PAP > 50 mmHg)
* cardiac failure or EF < 40% or intra-aortic balloon use
* pulmonary hypertension over 50 mmHg
* severe renal insufficiency
* history of allergy or intolerance to: morphine, acetaminophen, ropivacaine.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-04-27 (Actual); Primary Completion 2015-01-19 (Actual); Study Completion 2015-01-19 (Actual)

PRIMARY OUTCOMES:
The deadline for obtaining all criteria consistent with an output of postoperative intensive care | 72 hours
  The criteria will be considered by an independent adjudication committee unaware of the treatment given, according to a predefined checklist, whatever the actual delay for discharge. The checklist was built with the help of published recommendations [Camp et al. J Card Surg 2009; 24:414].

SECONDARY OUTCOMES:
Surgery time | 24 hours
Quantity of sufentanil administered | 72 hours
Total morphine consumption | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Vedat Eljezi, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Eljezi V, Imhoff E, Bourdeaux D, Pereira B, Farhat M, Schoeffler P, Azarnoush K, Duale C. Bilateral sternal infusion of ropivacaine and length of stay in ICU after cardiac surgery with increased respiratory risk: A randomised controlled trial. Eur J Anaesthesiol. 2017 Feb;34(2):56-65. doi: 10.1097/EJA.0000000000000564. PMID 27977439